#### STUDY PROTOCOL

# 1. Title of the Study

Clinical Profile of Appendicitis and Comparative Study of Harmonic Scalpel (Seal and Cut) Versus Suture Ligation of the Base of Appendix During Laparoscopic Appendectomy

# 2. Protocol ID & Registration

Protocol ID: GSVM/GENSURG/APP/2025

ClinicalTrials.gov Identifier (NCT Number): [To be added]

Trial Registration Registry: ClinicalTrials.gov

# 3. Principal Investigator

Name: Dr. Apoorva Mathur

Designation: Principal Investigator

Affiliation: Department of General Surgery, GSVM Medical College, Kanpur, India

Email:apoorvamathur05@gmail.com

Phone: 8484805719

# 4. Research Guide / Senior Author

Name: Dr. G.D Yadav

Designation: Professor & Head

Department: General Surgery, GSVM Medical College, Kanpur

## **5.** Background and Rationale

Acute appendicitis is a common surgical emergency. Laparoscopic appendectomy is widely accepted, with secure closure of the appendix base being a critical step. The harmonic scalpel offers an energy-based alternative to traditional suturing. This study aims to compare outcomes between these two techniques.

# 6. Study Objectives

Primary Objective:

- To compare operative time between harmonic scalpel and suture ligation techniques.

# Secondary Objectives:

- To evaluate postoperative complications (leak, ileus, SSI)
- To assess hospital stay duration
- To document appendix position intraoperatively

# 7. Study Design

Study Type: Interventional (Clinical Trial) Allocation: Randomized (computer-based) Interventional Model: Parallel Assignment Masking: Single (Participant)

Number of Arms: 2

Primary Purpose: Treatment

# 8. Participants

Sample Size: 60 patients (30 per group)

#### **Inclusion Criteria:**

- Age 15-60 years
- Diagnosed with uncomplicated acute appendicitis
- Consent to participate

#### **Exclusion Criteria:**

- Perforated/gangrenous appendix
- Pregnancy
- Coagulopathy or severe comorbid illness

## 9. Interventions

Arm A: Harmonic Scalpel Group (Experimental)

Laparoscopic appendectomy using harmonic scalpel to seal and divide appendix base.

Arm B: Suture Ligation Group (Active Comparator)

Laparoscopic appendectomy with intracorporeal suture ligation of appendix base.

#### 10. Outcome Measures

Primary Outcome:

- Operative time (in minutes)

#### **Secondary Outcomes:**

- Position of appendix (intraoperative)
- Postoperative leak (within 7 days)
- Postoperative ileus (within 3 days)
- Surgical site infection (within 30 days)
- Hospital stay (in days)

#### 11. Ethical Considerations

Approved by Institutional Ethics Committee, GSVM Medical College Informed written consent will be obtained from all participants Trial will be registered with ClinicalTrials.gov

## 12. Data Sharing Statement

De-identified individual data will be shared upon request for secondary analysis after 6 months of publication.

# 13. Timeline

Study Start: [April 2024]

Estimated Completion: [e.g., july 2025]

# **14. Funding and Support**

No external funding. Supported by institutional resources.

Date- 01/05/2025